CLINICAL TRIAL: NCT05297370
Title: Mixed and Match Versus One-size-fits-all: A Randomized Controlled Trial of Self-determination Theory on a Menu of Smoking Cessation Options (SDTM) Among Adult Smokers
Brief Title: Mixed and Match vs One-size-fits-all
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDTM-adult
Record Dates: First submitted 2021-05-18; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Smoking Cessation
Keywords: self-determination theory; adult smokers; Mixed and match; one-size-fits-all; feasibility; abstinence; quit
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed and Match (Other): Participants can choose to receive their own smoking cessation treatment options from our menu.
  Interventions: Behavioral: Mixed and match Intervention
- Control (Other): Participants will receive a self-help quitting leaflet
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Mixed and match Intervention — Participants will receive a brief 15-minute counselling session based on the 5A's' and '5R's' models by our trained research assistant. Participants will be able to choose their smoking cessation treatment options from our menu.
  Arms: Mixed and Match
Other: Control — Participants in the control group will receive a self-help quitting leaflet issued by the TACO
  Arms: Control

SUMMARY:
Most existing smoking cessation services are based on '5A's' and '5R's' models which are recognized by the World Health Organization as a standardized tool for smoking cessation. While there are more techniques that are known to be effective and could be incorporated in existing smoking cessation interventions to further promote their effectiveness. This study is to examine the effectiveness SDTM in assisting adult smokers in Hong Kong to quit.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will be conducted. One-hundred adult smokers aged 25 or above will be recruited from smoking hotspots in Hong Kong. Participants in the intervention group will be contacted by our trained research assistant to receive a telephone counselling session at baseline. Participants can choose to receive their own smoking cessation treatment options from our menu. Control group participants will only receive a self-help quitting leaflet

ELIGIBILITY:
Inclusion Criteria:

* have smoking in the previous 30 days.
* be above 25 years old
* able to speak Cantonese and read Chinese

Exclusion Criteria:

* who are receiving current smoking cessation services
* report psychological disorders
* at risk of suicide

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported abstinence at 6-month follow-up | At 6-month follow-up
  participants will be asked about their self-reported abstinence in the past 7 and 30 days
Biochemically validated abstinence | At 6 months follow-up
  validate the self-reported abstinence if the level of carbon monoxide in expired air was less than 4 parts per million and saliva cotinine level was less than100 ng/mL in parallel tests
Self-efficacy at 6-month follow-up | At 6-month follow-up
  Participants will be asked about their self-efficacy in quitting. The score ranges from 0 to 10. Higher scores represent a higher self-efficacy.

SECONDARY OUTCOMES:
Screening rate | at day 1
  calculated as the number of smokers screened at smoking hotspots by the RA divided by number of smokers available
Eligibility rate | at day 1
  calculated by dividing the number of smokers who are eligible by the number who are screened.
Randomization rate | at day 1
  calculated by dividing the number of smokers who are randomized into intervention and control groups by those who provide consent.
Attendance rate | Immediately after the training workshop
  calculated by dividing the number of smokers who complete the intervention by those who are randomized.
Retention rate at 1-week follow-up | At 1-week follow-up
  calculated by dividing the number of smokers who remain in the study by those who are randomized
Retention rate at 1-month follow-up | At 1-month follow-up
  calculated by dividing the number of smokers who remain in the study by those who are randomized
Retention rate at 6-month follow-up | At 6-month follow-up
  calculated by dividing the number of smokers who remain in the study by those who are randomized
Retention rate at 3-month follow-up | At 3-month follow-up
  calculated by dividing the number of smokers who remain in the study by those who are randomized
Adherence to intervention protocol at 1-week follow-up | At 1-week follow-up
  calculated by dividing the number of smokers who follow and practice the chosen treatment options by those who are randomized
Adherence to intervention protocol at 1-month follow-up | At 1-month follow-up
  calculated by dividing the number of smokers who follow and practice the chosen treatment options by those who are randomized
Adherence to intervention protocol at 3-month follow-up | At 3-month follow-up
  calculated by dividing the number of smokers who follow and practice the chosen treatment options by those who are randomized
Adherence to intervention protocol at 6-month follow-up | At 6-month follow-up
  calculated by dividing the number of smokers who follow and practice the chosen treatment options by those who are randomized
Complete rate at 1-week follow-up | At 1-week follow-up
  calculated by dividing the number of smokers who returned questionnaires by the number of questionnaires distributed
Complete rate at 1-month follow-up | At 1-month follow-up
  calculated by dividing the number of smokers who returned questionnaires by the number of questionnaires distributed
Complete rate at 3-month follow-up | At 3-month follow-up
  calculated by dividing the number of smokers who returned questionnaires by the number of questionnaires distributed
Complete rate at 6-month follow-up | At 6-month follow-up
  calculated by dividing the number of smokers who returned questionnaires by the number of questionnaires distributed
Missing data at 1-week follow-up | At 1-week follow-up
  calculated as the percentage of missing values in the dataset
Missing data at 1-month follow-up | At 1-month follow-up
  calculated as the percentage of missing values in the dataset
Missing data at 3-month follow-up | At 3-month follow-up
  calculated as the percentage of missing values in the dataset
Missing data at 6-month follow-up | At 6-month follow-up
  calculated as the percentage of missing values in the dataset
Adverse events at 6-month follow-up | At 6-month follow-up
  Participants will report any unfavorable and unintended events
Adverse events at 1-week follow-up | At 1-week follow-up
  Participants will report any unfavorable and unintended events
Adverse events at 1-month follow-up | At 1-month follow-up
  Participants will report any unfavorable and unintended events
Adverse events at 3-month follow-up | At 3-month follow-up
  Participants will report any unfavorable and unintended events
Self-reported abstinence at 1-week follow-up | At 1-week follow-up
  Participants will be asked about their self-reported abstinence in the past 7 and 30 days
Self-reported abstinence at 1-month follow-up | At 1-month follow-up
  participants will be asked about their self-reported abstinence in the past 7 and 30 days
Self-reported abstinence at 3-month follow-up | At 3-month follow-up
  participants will be asked about their self-reported abstinence in the past 7 and 30 days
Self-efficacy at 1-week follow-up | at 1-week follow-up
  Participants will be asked about their self-efficacy in quitting. The score ranges from 0 to 10. Higher scores represent a higher self-efficacy.
Self-efficacy at 1-month follow-up | at 1-month follow-up
  Participants will be asked about their self-efficacy in quitting. The score ranges from 0 to 10. Higher scores represent a higher self-efficacy.
Self-efficacy at 3-month follow-up | at 3-month follow-up
  Participants will be asked about their self-efficacy in quitting. The score ranges from 0 to 10. Higher scores represent a higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Lam, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No